CLINICAL TRIAL: NCT06568081
Title: SloMo2: A Process Evaluation, Effectiveness, and Cost-effectiveness Study of a Digitally Supported Therapy for Psychosis in Routine Care
Brief Title: SloMo2: Implementation, Effectiveness, and Cost-effectiveness Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Sussex Partnership NHS Foundation Trust (Other); Northumberland, Tyne and Wear NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 338439
Record Dates: First submitted 2024-08-13; First posted 2024-08-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Affective Psychoses
Keywords: Digital health; User-centred design
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Affective Disorders, Psychotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SloMo (Experimental)
  Interventions: Other: SloMo

INTERVENTIONS:
Other: SloMo — SloMo, is a blended digital therapeutic for people who fear harm from others. It is based on cognitive-behavioural therapy for psychosis. An online therapy platform supports the delivery of 11 face-to-face modules, which are synchronised to a native mobile app for use in daily life. SloMo works by helping people to notice their worries and fast thinking habits, and encourages them to slow down for a moment to find ways of feeling safer.

SUMMARY:
Worries about harm from others (also known as paranoia) are common. Thinking fast or going on gut feelings is natural but can fuel these worries. For some, fast thinking and worries start to get in the way of life. Cognitive behaviour therapy for psychosis (CBTp) is the recommended talking therapy. However, only a minority of people can access CBTp due to limited resources, and even when available, therapy can be difficult to do and use in daily life.

SloMo is a digitally supported therapy that aims to overcome these barriers, and was developed by people with psychosis, designers, and psychologists. It supports people to notice worries and fast thinking habits. During therapy sessions, people learn to slow down and feel safer. Personalised spinning thought bubbles are slowed down using SloMo tips. An app provides access to helpful messages.

SloMo was previously tested in a randomised trial of 361 people attending mental health services. SloMo was found to be safe to use, with no adverse events linked to the software. People in the SloMo group had lower paranoia, and better confidence and wellbeing, over 6 months compared to people who just received their usual care. People found SloMo enjoyable and easy to use.

The next step is to evaluate if SloMo can be safely and effectively delivered by therapists working in NHS services. If SloMo works in routine care, the therapy will be made more widely available in the NHS.

An improved version of SloMo has been co-produced based on feedback. Sixty therapists will be trained and supervised in 3 trusts to deliver SloMo to 150 people who fear harm from others. Safety, technical performance, uptake, engagement and acceptability data, alongside interviews with patients, therapists, and managers, will investigate how SloMo is used. Paranoia severity and wellbeing will be measured pre, post therapy, and at 12 months follow up, to find out if SloMo helps. Service use data will evaluate costs and savings.

DETAILED DESCRIPTION:
DESIGN AND AIMS The study is a repeated measures design, with clinical outcome assessments pre-, post-delivery of SloMoR2, and a 12-month follow-up. The aim is to evaluate if SloMo is implementable and effective when delivered in routine care by therapists working in NHS routine services. Delivery with high and low intensity therapists will be evaluated, with the former holding doctorate or diploma therapy qualifications, and the latter representing graduate psychologists or the NHS's expanding workforce of psychological practitioners. Outcomes will be evaluated using questionnaires, software analytics, and medical record data (for adverse events, service use, and demographics when not self-reported). Interviews will be conducted with a subgroup of relevant stakeholders to understand their experiences of SloMo.

The project will be conducted in 3 NHS trusts. Each trust will have a local study team, funded by the research grant and directly employed by local services, to support training, supervision, and implementation. Design research has already been conducted in preparation for the study to support the co-production of an improved version of SloMo tailored for implementation (SloMoR2). The study will run for 42 months and consists of four stages:

1. Site set-up (month 1-3) Site set-up will be conducted to pilot the training, supervision, and technical support procedures that will ensure SloMoR2's performance, data protection and clinical safety.

2a. Process evaluation: Implementation (month 4 - 39) A mixed-method process evaluation will be co-produced to understand how SloMoR2 is experienced, including safety, engagement, adherence, acceptability, fidelity & usability, and to identify barriers and enablers to implementation.

2ba. Effectiveness and cost-effectiveness (month 4 - 39) An evaluation will be conducted to establish the effectiveness and cost-effectiveness of SloMoR2 when delivered in routine care, including 12 month follow-up.

3. Analysis, resource development and dissemination (month 40 - 42) Findings will be summarised in consultation with our LEAP group. They will be written up in a plain English summary and as articles for submission to peer-review publications. Experiences of therapy delivery will inform any further refinements to the SloMoR2 software. Findings will also be used to support the co-design of an automated e-learning programme for therapists and develop a commercialisation strategy to assist being scaled up in the NHS.

SAMPLE AND RECRUITMENT Service user recruitment: The recruitment target is to deliver SloMo to 150 service user participants (across Stage 1 and 2) who are: Aged ≥18 years, meet criteria for ICD-10 psychosis diagnoses (F20-29, F30-39), seeking therapy for paranoia, in contact with secondary care mental health services, and capable of providing informed consent to engage in therapy. People will be excluded if they: are at acute risk of harm to self or others, are unable to engage in therapy due to language barriers, and have a primary diagnosis of alcohol/substance dependence, learning disability, or organic brain injury or illness implicated in psychosis.

Therapist recruitment, training, and supervision: In Stage 1, an initial cohort of therapists ('high intensity'; n = 5 per trust) will be selected from senior clinicians experienced in delivery and supervision of CBT for psychosis. Therapists will be required to complete a 1-day training. They will subsequently be able to access on-demand clinical and technical supervision from their local study team as required to support SloMoR2 delivery. In Stage 2, a further 45 'high' and 'low' intensity therapists will be trained across the 3 sites. Training will be extended to 3 days for low intensity therapists. The local study team will liaise with local services to promote SloMo2 and support trainers to roll out training to other high and low intensity therapists.

Stakeholder recruitment: The experience of SloMo's delivery will be evaluated using subgroups of the therapist and participant samples recruited in Stages 1 and 2 (N = 60, and N = 150, respectively). This will involve interviewing subgroups of service users (n = 20) and therapists (n = 6) involved in SloMo's delivery, as well as senior managers (n = 5) and payers (stakeholders involved in the commissioning of mental health services; n = 5), about their experience of SloMo. The service users will be recruited by the local study team, and will be invited to interview post-therapy and at 12-month follow-up. The team will approach participants who consented to be contacted about further SloMo studies, once the participant has disengaged (therapist defined) or completed therapy. The four samples will be recruited to ensure a diverse range with respect to age, ethnicity, gender, site, and professional background (for staff interviews). All potential participants will be provided with a participant information sheet and given the opportunity to ask questions before signing the consent form.

PROCEDURE The local study team will initially conduct PPI consultation with their trust therapy workforce to scope readiness for adoption of SloMoR2. This work will identify implementation barriers and facilitators, to enable tailoring of implementation resources and strategies to site needs.

Trained therapists will identify potential participants and offer them SloMo, based on their clinical judgement. Following an initial introduction, participants will provide informed consent to receive SloMo and for their data to be collected for research purposes, with an optional opt-in for contact about further SloMo research. The burden of the informed consent process will be minimised where possible. This has been done by embedding the participant information sheet and consent form at the beginning of the SloMo webapp ('therapy platform'). Therapists will review this with potential participants and address any questions they have. Data storage and strategies for data protection will be emphasised, based on PPI feedback that this is a key area of concern. It will also be emphasised that service users will be free to withdraw their consent to engage in therapy at any time or to request that their data be deleted from the SloMo software or omitted from the research analysis.

If willing to proceed, participants' consent will be provided by indicating consent on the form. Participants will not sign the consent form with their name, to minimise the personally identifiable information stored in the software. Therapists will countersign and date the consent form. A copy of the countersigned consent form will be posted or sent electronically to the participant by the local SloMo team.

Pre and post therapy measures will be collected through the SloMo therapy platform at the first (R-GPTS (part B), short WEMWBS), second (GBO) and last therapy session (all), and will be repeated at 12-months post-consent. Sessional measures will be taken at each session and at 12-months follow-up. The local study team will collect demographic information from participants directly, and will extract adverse event and service use data from participants' medical record.

INTERVENTION SloMoR2 consists of up to 11 digitally supported therapy platform modules targeting paranoia and a mobile app for use outside of sessions. Therapy will be delivered according to the SloMo manual instructions for use. The therapy helps people learn to slow down for a moment to find ways of feeling safer and living well. Animated stories and interactive tasks support participants to learn how to apply SloMo tips to manage their worries, with in-session content synchronised to the mobile app which provides out of session support.

OUTCOMES

1a) Implementation To address the primary research question, is SloMoR2 implementable in routine care post-therapy, quantitative data will be gathered for the following primary outcomes: i) safety, measured by frequency of any unanticipated serious therapy and/or device-related adverse events, and ii) service user engagement, measured by the proportion of participants who are delivered 5 or more SloMo sessions ('minimum therapeutic dose'). In addition, data will be gathered for the following secondary outcomes: i) service user engagement, measured by the number of individuals who begin (1 or more sessions) and complete therapy (8 or more sessions, 'full course' as three modules are optional), ii) therapist uptake, measured by the percentage of therapists that receive SloMo R2 training who commence therapy with at least one participant, iii) adherence, measured by percentage completion of sessions started, iv) usage, service user usage of mobile app, v) acceptability, measured by the percentage of positive responses on the NHS Family and Friends Test, vi) fidelity, competence of therapy delivery (with a random selection of 10 sessions per site assessed by the local study lead), vii) stakeholder experience of implementation, based on qualitative interviews with service users, therapists, senior managers, and payers, and viii) usability, measured by the User Experience Survey (UES; Service user and therapist).

To address the secondary research question, is SloMoR2 implementable in routine care at 12-month, quantitative safety data and qualitative data regarding stakeholder experiences will also be gathered to 12-month follow up.

The qualitative interviews exploring user experience in participants who have been offered SloMo will be lived experience researcher-led. The qualitative interviews with therapists will explore experiences of training and delivery of SloMoR2 in more detail. Finally, senior managers and payers, who have and have not been involved in implementing SloMo, will be interviewed to understand their perspective on SloMo and its scale-up. All interviews will be audio recorded and transcribed for analysis. Participants will be reimbursed for their time according to INVOLVE guidelines.

1b) Effectiveness To address the primary research question, is SloMoR2 effective for paranoia and wellbeing when delivered in routine care post-therapy, participants will complete (via the SloMo therapy platform) three brief questionnaires at the beginning and end of therapy. The primary effectiveness outcome measure is the persecution subscale (part B) of the Revised Green Paranoid Thoughts Scale (RGPTS-B). Secondary effectiveness outcome measures are the short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) and the Goal Based Outcome Scale. Sessional measures will be collected during therapy sessions to monitor progress, using four scales (rated from 0 - 100) of paranoia distress, fast and slow thinking, safety beliefs and confidence. To address the secondary research question, is SloMoR2 effective for paranoia and wellbeing when delivered in routine care at 12-months follow-up, participants will re-complete the RGPTS-B, SWEMWBS, GBOS and sessional measures.

1b) Cost-effectiveness To address the primary research question, is SloMoR2 cost-effective when delivered in routine care, costs and savings will be evaluated by the local study team extracting mental health service use data from participant medical records using the Client Service Receipt Inventory (CSRI), and QALYs derived from an algorithm applied to the Revised Green Paranoid Thoughts Scale, persecution subscale (part B) (RGPTS-B). Mental health service use data will cover the 6-month period prior to the intervention, and a 12-month period following consent (including both the intervention period and follow-up). This analysis will also incorporate the service use data collected for the SlowMoR1 trial as this will provide additional data to enhance the health economic modelling.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for ICD-10 psychosis diagnoses (F20-29, F30-39)
* Seeking therapy for paranoia
* In contact with secondary care mental health services
* Capacity to provide informed consent to engage in therapy

Exclusion Criteria:

* Acute risk of harm to self or others
* Unable to engage in therapy due to language barriers
* Primary diagnosis of alcohol/substance dependence, learning disability, or organic brain injury or illness implicated in psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Implementation: Safety (adverse event incidence) | Pre-therapy to post-therapy.
  Frequency of any unanticipated serious therapy and/or device-related adverse events
Implementation: Service user engagement | Duration of therapy (typically up to 6 months)
  Proportion of participants who are delivered 5 or more SloMo sessions ('minimum therapeutic dose')
Effectiveness: Paranoid thoughts | Pre- to post-therapy.
  Revised Green Paranoid Thoughts Scale, persecution subscale (part B) (RGPTS-B, Freeman et al, 2021). Range 0-40, higher scores indicate worse outcome.
Cost-effectiveness: Service use | Pre-therapy to post-therapy.
  Unit costs calculated from the Client Service Receipt Inventory (CSRI, Beecham and Knapp, 2001)
Cost-effectiveness: Paranoid thoughts | Pre-therapy to post-therapy.
  QALYs derived from an algorithm applied to the Revised Green Paranoid Thoughts Scale, persecution subscale (part B) (RGPTS-B, Freeman et al, 2021)

SECONDARY OUTCOMES:
Implementation: Service user engagement | Duration of therapy (typically up to 6 months)
  Number of individuals who begin (1 or more sessions) and complete therapy (8 or more sessions, 'full course' as three modules are optional)
Implementation: Therapist uptake | Duration of study (42 months)
  Percentage of therapists that receive SloMo R2 training who commence therapy with at least one participant
Implementation: Adherence | Duration of therapy (typically up to 6 months)
  Percentage completion of sessions started.
Implementation: Usage | Pre- to post-therapy (typically up to 6 months)
  Percentage of service users meeting mobile app adherence criteria (at least 1 home screen interaction after a minimum of 3 therapy sessions).
Implementation: Acceptability | Post-therapy (typically up to 6 months)
  Percentage of positive responses on the NHS Family and Friends Test
Implementation: Fidelity | Duration of study (42 months)
  Proportion of therapists meeting competence on the Revised Cognitive Therapy Scale (CTS-R) (of a random selection of 10 sessions scored per site, assessed by the local study lead).
Effectiveness: Paranoid thoughts - follow-up | Pre-therapy to 12 months follow-up
  Revised Green Paranoid Thoughts Scale, persecution subscale (part B) (RGPTS-B, Freeman et al, 2021). Range 0-40, higher scores indicate worse outcome.
Cost-effectiveness: Paranoid thoughts - follow-up | Pre-therapy to 12 months follow-up.
  QALYs derived from an algorithm applied to the Revised Green Paranoid Thoughts Scale, persecution subscale (part B) (RGPTS-B, Freeman et al, 2021)
Cost-effectiveness: Service use - follow-up | Pre-therapy to 12 months follow-up.
  Unit costs calculated from the Client Service Receipt Inventory (CSRI, Beecham and Knapp, 2001)
Implementation: Safety (adverse event incidence) - follow-up | Pre-therapy to 12 months follow-up
  Frequency of any unanticipated serious therapy and/or device-related adverse events
Implementation: Stakeholder experience of implementation | Duration of study (42 months)
  Qualitative interviews with i) service users, ii) therapists, iii) senior managers, iv) payers
Implementation: Usability | Post-therapy (typically up to 6 months)
  User Experience Survey (UES, Hardy et al, 2022; Service user and therapist)
Effectiveness: Wellbeing | Pre- to post-therapy (typically up to 6 months)
  Short-Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, Stewart-Brown et al, 2009). Range 7-35, higher scores indicate better outcome.
Effectiveness: Sessional measures | Duration of therapy (typically up to 6 months)
  Collected using visual analogue scales (rated from 0 - 100) of paranoia distress, fast and slow thinking, safety beliefs and confidence
Effectiveness: Goal attainment | Pre- to post-therapy (typically up to 6 months)
  Goal Based Outcome (GBO, Law et al, 2015). Range 0 (no progress) to 10 (goal has been reached), higher scores indicate better outcome.
Effectiveness: Wellbeing - follow-up | Pre-therapy to 12 months follow-up
  Short-Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, Stewart-Brown et al, 2009). Range 7-35, higher scores indicate better outcome.
Effectiveness: Sessional measures - follow-up | Pre-therapy to 12 month follow-up
  Collected using visual analogue scales (rated from 0 - 100) of paranoia distress, fast and slow thinking, safety beliefs and confidence
Effectiveness: Goal attainment - follow-up | Pre-therapy to 12 months follow-up
  Goal Based Outcome (GBO, Law et al, 2015). Range 0 (no progress) to 10 (goal has been reached), higher scores indicate better outcome.
Cost-effectiveness: Wellbeing | Pre- to 6 months post-therapy.
  QALYs derived from an algorithm applied to the Short-Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, Stewart-Brown et al, 2009)
Cost-effectiveness: Wellbeing - follow-up | Pre-therapy to 12 months follow-up.
  QALYs derived from an algorithm applied to the Short-Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, Stewart-Brown et al, 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hardy, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A fully anonymised, aggregate dataset will be shared with the wider research community. We will upload the data resulting from the study to ClinicalStudyDataRequest.com (CSDR), a consortium of clinical study sponsors/funders which is endorsed by Wellcome. In addition, other researchers may request access to IPD by contacting the study team, and will be shared in line with access criteria below.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available after completion of data collection and analysis, and publication of the main outcome papers, and will be available indefinitely via CSDR.
Access Criteria: CSDR provides an ongoing forum where research proposals are checked and reviewed in 3 stages: 1) by the Wellcome Trust, which is the secretariat for the Independent Review Panel (IRP), 2) study funders sponsors and 3) the IRP.
  Direct requests for access must be accompanied by a protocol setting out the aims of the study for which the data are requested, very brief details of the credentials of team conducting the study (institutional affiliation, degrees or qualifications), methods outlined and appropriate ethical approval in place.